CLINICAL TRIAL: NCT01733017
Title: Nutrition Intervention to Reduce Symptoms in Patients With Advanced Heart Failure
Brief Title: Nutrition Intervention to Decrease Symptoms in Patients With Heart Failure
Acronym: NIHFT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Terry Lennie (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor-Investigator, Terry Lennie, PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01NR013430 (NIH)
Record Dates: First submitted 2012-11-15; First posted 2012-11-26 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Heart Failure
Keywords: heart failure; nutrition therapy; symptoms; quality of life; lycopene; omega-3 fatty acids
MeSH Terms: conditions — Heart Failure | interventions — Docosahexaenoic Acids; Rice Bran Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sodium reduction, omega-3, lycopene (Experimental): combination of dietary sodium restriction with supplementation of omega-3 capsules and lycopene containing juices or foods
  Interventions: Behavioral: Sodium reduction; Dietary Supplement: omega 3 and lycopene supplements
- Control (Placebo Comparator): Limited nutritional counseling, juice without lycopene, rice oil capsules
  Interventions: Dietary Supplement: rice bran oil capsules; Behavioral: Generic dietary feedback from

INTERVENTIONS:
Behavioral: Sodium reduction — Teaching and skill building to reduce dietary sodium
  Arms: sodium reduction, omega-3, lycopene
Dietary Supplement: omega 3 and lycopene supplements — omega-3 fatty acid supplements and juices containing lycopene
  Arms: sodium reduction, omega-3, lycopene
Dietary Supplement: rice bran oil capsules — placebo capsules
  Other Names: placebo
  Arms: Control
Behavioral: Generic dietary feedback from — Provided a summary of the 3 day dietary recalls at baseline, 3 months, and 6 months
  Other Names: attention control
  Arms: Control

SUMMARY:
The purpose of is to test the effects of a 6-month nutrition intervention of dietary sodium reduction combined with supplementation of lycopene and omega-3 fatty acids on heart failure symptoms, health-related quality of life, and time to heart failure rehospitalization or all-cause death.

DETAILED DESCRIPTION:
For a majority of patients with advanced heart failure, medical treatment is only partially effective in relieving heart failure symptoms. Therefore, it is recommended that palliative care be initiated soon after diagnosis. There is a need for complementary, nonpharmacologic interventions that could be easily implemented by health care providers to provide palliative care. Three major pathologic pathways underlying heart failure symptoms have been identified: fluid overload, inflammation, and oxidative stress. Prior research has demonstrated that three nutrients-sodium, omega-3 fatty acids, and lycopene-can alter these pathologic pathways. Clinical trials to date have only tested each nutrient individually. There is strong theoretical rationale that a combined intervention targeting all three nutrients would have substantial benefit in relieving symptoms in advanced heart failure. Therefore, the purposes of this study are to test the effects of a 6-month nutrition intervention of dietary sodium reduction combined with supplementation of lycopene and omega-3 fatty acids on heart failure symptoms, health-related quality of life, and time to heart failure rehospitalization or all-cause death. The aims of this placebo controlled study are 1) to determine the effects of a 6-month nutrition intervention on symptom burden (edema, shortness of air, and fatigue) and health related quality of life at 3 and 6 months, and time to heart failure rehospitalization or all-cause death over 12 months from baseline; 2) compare dietary sodium intake, inflammation, and markers of oxidative stress between the nutrition intervention group and a placebo group at 3 and 6 months; and 3) compare body weight, serum lycopene, and erythrocyte omega-3 index between the nutrition intervention group and a placebo group at 3 and 6 months. A total of 150 patients with advanced heart failure will be randomized to either the nutrition intervention or placebo group (75 per group). The nutrition intervention group will receive a theory based education and skill building intervention designed to decrease dietary sodium intake to ~2 g per day. A research nurse will make 4 home visits and one follow-up telephone call over 6 months to provide the education-skill building intervention. The intervention group will take 3 omega-3 fatty acid capsules (350 mg eicosapentaenoic acid and 50 mg docosahexaenoic acid) and consume tomato juice or other tomato-based products containing 20-25 mg of lycopene daily for six months. The placebo group will receive the same number of visits and phone calls but only general nutrition information will be provided. They will take 3 placebo capsules containing rice oil (500 mg/capsule) and consume their choice of fruit juices that do not contain lycopene daily for six months. Data will be collected in person at baseline, 3 months, and 6 months by a research assistant blinded to the group assignment. Patients will be followed for an additional 6 months by telephone to collect longer term data on symptom burden and quality of life as well as heart failure hospitalization and all-cause mortality at 9 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* chronic heart failure with either preserved or non-preserved ejection fraction
* for chronic heart failure, have undergone evaluation of heart failure and optimization of medical therapy, for patients discharged from hospital for acute/newly diagnosed heart failure, have undergone evaluation of heart failure and optimization of medical therapy for at least 1 month post discharge
* New York Heart Association functional classification of II, III or IV
* have not been referred for heart transplantation
* able to read and speak English
* no cognitive impairment that precludes giving informed consent or ability to follow protocol instruction.

Exclusion Criteria:

* BMI < 17 kg/m2 or > 46 kg/m2
* co-existing illness documented in the medical record known to be associated with systemic inflammation decreased appetite or absorption, fatigue, edema, or weight loss
* currently taking dietary supplements that contain lycopene or omega-3 fatty acids
* allergy to rice bran oil

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-11; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Event-Free Survival | 12 months
  Combined endpoint of cardiac-related hospitalization and all cause mortality
Symptom burden | baseline, 3, 6, 9, and 12 months
  combined score of symptom severity, frequency, and distress for common symptoms of heart failure
Quality of life | baseline, 3, 6, 9, 12 months
  heart failure related quality of life

SECONDARY OUTCOMES:
omega-3 index | baseline, 3, 6, 9, 12 months
  the ratio of EPA plus DHA as a percentage of total fatty acids in the cell membrane of erythrocytes
oxidative stress | baseline, 3, 6, 9, 12 months
  serum levels of malondialdehyde and 8-iso-PGF2a isoprostane will serve as markers of increased lipid peroxidation due to oxygen free radical production exceeding antioxidant capacity
Inflammation | baseline, 3, 6, 9, 12 months
  Serum levels of tumor necrosis factor-alpha (TNFα), soluble TNF receptors: sTNFR1 and sTNFR2 will be measured as markers of proinflammatory cytokine activity; interleukin-10 (IL-10) will be measured as a marker of anti-inflammatory cytokine activity
Lycopene | baseline, 3, 6, 9, 12 months
  Plasma lycopene will be measured as a marker intervention effectiveness
Sodium intake | baseline, 3, 6, 9, 12 months
  Three 24-hour diet recall interviews at each timepoint will be used estimate sodium intake and to identify high sodium foods and eating patterns for the sodium reduction component of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Terry A Lennie, PhD, Principal Investigator — University of Kentucky College of Nursing
Locations (2):
- United States (2):
  - University of Kentucky, College of Nursing, Lexington, Kentucky
  - Norton Health Care, Louisville, Kentucky